CLINICAL TRIAL: NCT04100304
Title: Preoperative Evaluation of the Remaining Part of the Liver for Liver Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moaz Ahmed Sayed Ahmed, resident doctor at general surgery department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: liver resection
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient under going liver resection (Other)
  Interventions: Diagnostic Test: resection

INTERVENTIONS:
Diagnostic Test: resection — CT volumetry,liver function,biopsy before resection

SUMMARY:
* Review the outcomes of the current treatments modalities.
* Give an effective treatment .
* Improve the outcome of these patients and decease rate of recurrence and complications.
* An adequate future liver remnant (FLR) reduces the risk of postoperative liver failure after major hepatectomy.
* incurs a risk of postoperative liver dysfunction and infection and there is a lack of objective evidence relating residual liver volume to these complications

DETAILED DESCRIPTION:
A liver resection is the surgical removal of all or a portion of the liver. It is also referred to as a hepatectomy, full or partial. A complete liver resection is performed in the setting of a transplant a diseased liver is removed from a deceased donor (cadaver). A living donor may also provide a piece of liver tissue which is procured through a partial hepatectomy, The procedure may be performed through a traditional open procedure or using minimally invasive techniques.

When is Liver Resection Performed Most hepatectomies are performed for the treatment of hepatic neoplasms, both benign or malignant. Benign neoplasms include hepatocellular adenoma, hepatic hemangioma and focal nodular hyperplasia.The most common malignant neoplasms (cancers) of the liver are metastases; those arising from colorectal cancer are among the most common, and the most amenable to surgical resection. The most common primary malignant tumour of the liver is the hepatocellular carcinoma. Hepatectomy may also be the procedure of choice to treat intrahepatic gallstones or parasitic cysts of the liver.

Liver surgery is safe when performed by experienced surgeons with appropriate technological and institutional support. As with most major surgical procedures, there is a marked tendency towards optimal results at the hands of surgeons with high caseloads in selected centres (typically cancer academic medical centers and transplantation centers).

Partial hepatectomy is surgery to remove part of the liver. Only people with good liver function who are healthy enough for surgery and who have a single tumor that has not grown into blood vessels can have this operation.

Imaging tests, such as CT or MRI with angiography are done first to see if the cancer can be removed completely. Still, sometimes during surgery the cancer is found to be too large or has spread too far to be removed, and the surgery that has been planned cannot be done.

Can a portion of the remaining normal liver grow back? When a portion of a normal liver is removed, the remaining liver can grow back (regenerate) to the original size within several weeks. A cirrhotic liver, however, cannot grow back. Therefore, before resection is performed for HCC, the non-tumor portion of the liver should be biopsied to determine whether there is associated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver resection for benign or malignant hepatic neoplasm at the time of study(two years)
* Patient consent.
* Age of the patient : Any age

Exclusion Criteria:

* patients has contraindication to do liver resection surgery.
* patients who are unfit for any surgical interventions.
* patients who refuse the operation or refusing to share his data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation | preoperative
  Evaluation of the remaining part of the liver by CTvolumetry for further management as liver transplant

SECONDARY OUTCOMES:
energy expenditure | [ Time Frame: 30 days ]
  Change in total energy expenditure (Kcal) following liver resection
Procedural parameters | intraoperative
  including intraoperative blood loss
Long-term outcomes | 5 years
  5-year tumor recurrence rate
Perioperative liver function | 30 days preoperative
  including serum levels of alanine aminotransferase (ALT)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang Z, Sun H, Li K, Yao W, Dong K, Ma Y, Zheng S. Prognostic factor analysis of stage 4S neuroblastoma in infant patients: A single center study. J Pediatr Surg. 2019 Dec;54(12):2585-2588. doi: 10.1016/j.jpedsurg.2019.08.031. Epub 2019 Aug 30. PMID 31521373
- [Background] Horiuchi T, Haruki K, Shiba H, Sakamoto T, Saito N, Shirai Y, Iwase R, Fujiwara Y, Yanaga K. Assessment of Outcome of Hepatic Resection for Extremely Elderly Patients With a Hepatic Malignancy. Anticancer Res. 2019 Sep;39(9):5143-5148. doi: 10.21873/anticanres.13709. PMID 31519626 (Retraction: PMID 31704878 Anticancer Res. 2019 Nov;39(11):6418)
- [Background] Rotellar F, Marti-Cruchaga P, Zozaya G, Tuero C, Lujan J, Benito A, Hidalgo F, Lopez-Olaondo L, Pardo F. Standardized laparoscopic central hepatectomy based on hilar caudal view and root approach of the right hepatic vein. J Hepatobiliary Pancreat Sci. 2020 Jan;27(1):E7-E8. doi: 10.1002/jhbp.669. Epub 2019 Oct 10. PMID 31518491
- [Background] Huiskens J, Bolhuis K, Engelbrecht MR, De Jong KP, Kazemier G, Liem MS, Verhoef C, de Wilt JH, Punt CJ, van Gulik TM; Dutch Colorectal Cancer Group. Outcomes of Resectability Assessment of the Dutch Colorectal Cancer Group Liver Metastases Expert Panel. J Am Coll Surg. 2019 Dec;229(6):523-532.e2. doi: 10.1016/j.jamcollsurg.2019.08.1445. Epub 2019 Sep 11. PMID 31520695